CLINICAL TRIAL: NCT04638907
Title: Fine Tuning of Deep Neuro-muscular Blockade in Robot-assisted Urological Surgery: A Prospective Proof of Concept Investigation
Brief Title: Fine Tuning of Neuro-muscular Blockade in Robot-assisted Prostatectomy
Acronym: NMBUro
Status: Completed | Type: Observational
Sponsor: Peter Biro (Other)
Responsible Party: Sponsor-Investigator, Peter Biro, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC ID 2016-01781
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Maintenance of Deep NM Block Without Overdosing
Keywords: neuromuscular block, robot-assisted prostatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational study group: Consenting adult male patients undergoing elective robot-assisted prostatectomy. No further selection or randomisation. Enrollment as availability for the study.
  Interventions: Procedure: Assessment of NM block

INTERVENTIONS:
Procedure: Assessment of NM block — Observation of resulting course of NM block under teratment and monitoring as described.

SUMMARY:
Assessing the routinely used protokoll for deep NM Block during robot-assisted prostatectomy in general anesthesia. The protocoll contains the repeated dosing of rocuronium according to the results of relaxometry performed with a TOFcuff relaxometer (RGB Medical, Madrid) during pneumoperitoneum. This is done by keeping the block level between 1 to 6 PTC (post tetanic counts). The scope of the study was to find out, to which percentage this protocoll permits the maintenance of block level inside of the desired range.

DETAILED DESCRIPTION:
Robot-assisted urological interventions require sufficiently deep neuromuscular relaxation (NMR) during the phase of pneumoperitoneum. This is achieved by repeated administration of the non-depolarizing neuromuscular relaxant rocuronium, which is used in clinical routine. The level of relaxation is usually measured with the TOF-Watch relaxometer. This device has limitations in its usability and accuracy in this setting because it is unreliable when the monitored arm of the patient is not accessible for the anaesthetist for visual or tactile assessment of finger movements. The novel TOF-Cuff relaxometry equipment is by design intended to provide constant and reliable quantitative and in vivo calibrated relaxometric values independently of the arm position. The combination of frequently adjusted neuromuscular relaxation in a standardised mode in combination with a reliable relaxometry by TOFcuff promises an improved surveillance of neuromuscular relaxation and a higher safety standard. This investigation aims to test and to define the combined use of the best available drug with the best available relaxometer for general anesthesia in robot-assisted urological surgery.

ELIGIBILITY:
Inclusion Criteria:

* consenting male adults undergoing elective robot-assisted urological surgery.

Exclusion Criteria:

* Emergency cases, Patients who don't understand the requirements of the study and don't agree to sign the informed consent. Contraindication to neuromuscular relaxation with rocuronium.

Ages: 18 Years to 90 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men have prostatectomy.
Study Population: Unselected pateints, who fulfil the inclusion criteria as they become available for anesthesia and surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Successful deep NM block | Entire duration of pneumoperitoneum varying between 2 and 5 hours.
  Time percentage of optimal NM block during pneumoperitoneum

SECONDARY OUTCOMES:
Surgeon's satisfaction | Duration of pneumoperitoneum
  Overall subjective satisfaction with the patient's relaxation by the surgeon on a verbal rating scale (1 = extremely bad; 10 = excellent)(Staehr-Rye 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, Prof. Dr., Study Chair — Institute of Anesthesiology, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Institue of Anesthesiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan to share the obtained data.